CLINICAL TRIAL: NCT03437278
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2b Dose-finding Study to Investigate the Efficacy and Safety of Ligelizumab (QGE031) in Adolescent Patients With Chronic Spontaneous Urticaria (CSU)
Brief Title: Study to Investigate the Efficacy and Safety of QGE031 in Adolescent Patients With Chronic Spontaneous Urticaria (CSU)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQGE031C2202; 2017-004207-52 (EudraCT Number)
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Anti-IgE; Chronic spontaneous urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — ligelizumab

STUDY DESIGN:
Intervention Model Description: This was a Phase 2b dose-finding, randomized, double-blind, parallel group, placebo controlled multicenter study in adolescent patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigator staff and personnel performing the study assessments remained blinded to the identity of the treatment from the time of randomization until final database lock. Data managers, programmers, statisticians, pharmacometricians and clinical experts of the Novartis trial team also remained blinded until final database lock. The study drug was prepared by an independent unblinded pharmacist (or authorized delegate) and administered by an independent unblinded administrator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ligelizumab 120 mg (Experimental): Participants received a dose of ligelizumab 120 mg (high dose) which consisted of one injection of 1 ml of ligelizumab 120 mg/ 1 ml vial every 4 weeks from Day 1 to Week 20 (inclusive).
  Interventions: Drug: Ligelizumab
- Ligelizumab 24 mg (Experimental): Participants received a dose of ligelizumab 24 mg (low dose) which consisted of one injection of 0.2 ml of ligelizumab 120 mg/ 1 ml vial every 4 weeks from Day 1 to Week 20 (inclusive).
  Interventions: Drug: Ligelizumab
- Placebo + Ligelizumab 120 mg (Placebo Comparator): Participants received Placebo which consisted of one injection of 1 ml placebo every 4 weeks from Day 1 to Week 8 (inclusive). From week 12 to week 20 (inclusive), participants received a dose of ligelizumab 120 mg (high dose) which consisted of one injection of 1 ml of ligelizumab 120 mg/ 1 ml vial.
  Interventions: Drug: Ligelizumab; Drug: Placebo

INTERVENTIONS:
Drug: Ligelizumab — Ligelizumab comes in 120 mg per 1 ml liquid vials. Participants received one injection every 4 weeks at a dose of 120 mg or 24 mg, high and low doses respectively.
  Other Names: QGE031
Drug: Placebo — Placebo 0 mg per 1 ml liquid injection once every 4 weeks.
  Arms: Placebo + Ligelizumab 120 mg

SUMMARY:
This clinical study was designed to evaluate the pharmacokinetics, safety and efficacy of ligelizumab in children from 12 to < 18 years of age, with chronic spontaneous urticaria (CSU). The participants were treated with ligelizumab as an add-on therapy to approved doses of H1 antihistamines (H1AH) following the guideline on treatment of CSU.

DETAILED DESCRIPTION:
This was a Phase IIb dose-finding, randomized, double-blind, parallel-group, placebo-controlled, multicenter study in adolescent patients. The study consisted of 3 distinct study periods: Screening, Treatment and Follow-up period.

After the screening period (up to 4 weeks), at Day 1 participants were randomized into one of the three treatment arms in 1:2:1 fashion to ligelizumab high dose (120 mg every four weeks (q4w)) versus ligelizumab low dose (24 mg q4w) versus placebo. During the 24 weeks of treatment period, doses were administered on Day 1 then on weeks 4, 8, 12, 16, and 20 weeks after randomization. Participants randomized to placebo received placebo on Day 1, Weeks 4 and 8; thereafter they received 120 mg ligelizumab (high dose) on Weeks 12, 16 and 20 such that by the end of the study, the same number of participants received ligelizumab high dose as low dose. The treatment period was followed by a treatment-free follow-up period of 16 weeks to a maximum of Week 40.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian's written informed consent and child's assent, if appropriate, must be obtained before any study related activity or assessment is performed. Of note, if the subject reaches age of consent (age as per local law) during the study, they will also need to sign the corresponding study ICF (Informed Consent Form) at the next study visit.
* Male and female adolescent patients aged ≥ 12 to <18 years at the time of screening.
* Diagnosis of CSU refractory to approved doses of H1-antihistamines at the time of randomization, as defined by all of the following:

  * The presence of itch and hives for at least 6 consecutive weeks at any time prior to enrollment despite current use of non-sedating H1-antihistamines during this time period
  * UAS7 score (range 0 - 42) ≥ 16 and HSS7 (range 0 - 21) ≥ 8 during 7 days prior to randomization (Day 1)
  * In-clinic UAS ≥ 4 on at least one of the screening visit days or Day 1 or a medical record of the presence of hives (confirmed and documented by a physician); patients must have been on H1-antihistamines for treatment of CSU at the time of in-clinic UAS at screening visit and/or time of the medical record of hives (for at least 3 days prior to the in-clinic UAS or medical record) • Patients must have been on H1-antihistamines for treatment of CSU for at least the 3 consecutive days immediately prior to the first screening visit and must have documented current use on the day of the initial screening visit
  * CSU diagnosis for ≥ 6 months
* Willing and able to complete a daily symptom e-Diary for the duration of the study and adhere to the study visit schedules.
* Demonstration of compliance with the e-Diary: patients should not have had any missing e-Diary entries in the 7 days prior to randomization. Re-screening may be considered.

Exclusion Criteria:

* Clearly defined underlying etiology for chronic urticarias other than CSU. This includes the following:

  * Inducible urticaria: urticaria factitia, cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic-, or contact-urticaria
  * Diseases with possible symptoms of urticaria or angioedema such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa), and hereditary or acquired angioedema (e.g., due to C1 inhibitor deficiency)
* Any other skin disease associated with chronic itching that might confound the study evaluations and results (e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis etc.)
* Previous exposure to omalizumab
* History of anaphylaxis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Argentina (3):
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Bahía Blanca
  - Novartis Investigative Site, Buenos Aires
- Novartis Investigative Site, Brussels, Belgium
- Canada (2):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Budapest, HUN, Hungary
- India (3):
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
- Russia (2):
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
- Spain (2):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
- Novartis Investigative Site, Taipei, Taiwan, Taiwan
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Aydin, Turkey
  - Novartis Investigative Site, Ankara

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Staubach P, Alvaro-Lozano M, Sekerel BE, Maurer M, Ben-Shoshan M, Porter M, Hua E, Ji Y, Burciu A, Savelieva M, Severin T, Drollmann A, Bienczak A. Ligelizumab in adolescents with chronic spontaneous urticaria: Results of a dedicated phase 2b randomized clinical trial supported with pharmacometric analysis. Pediatr Allergy Immunol. 2023 Jul;34(7):e13982. doi: 10.1111/pai.13982. PMID 37492920
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=985
- See also: A Pediatric Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 20 sites: Argentina (3), Belgium (1), Canada (2), Germany (2), Hungary (1), India (3), Russia (3), Spain (2), Taiwan (1) and Turkey (2).
Pre-assignment Details: Participants underwent a Screening period of up to 4 weeks.
Period: Overall Study
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Started | 24 | 13 | 12
Completed | 22 | 13 | 10
Not Completed | 2 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Progressive disease | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg | Total
Number analyzed (Participants) | 24 | 13 | 12 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.9 (1.94) | 15.2 (1.41) | 14.4 (1.51) | 14.8 (1.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 9 | 28
  Male | 14 | 4 | 3 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 1 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 16 | 12 | 10 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Weekly Urticaria Activity Score (UAS7) at Week 24
Description: UAS7 is a self-reported scoring system to evaluate urticaria signs and symptoms. UAS7 is the sum of daily urticaria activity scores (UAS) over a seven-day period. The possible range of UAS7 score is 0 to 42 (0 to 6 for daily UAS x 7 days). A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement. Baseline was calculated using data from the 7 days prior to the first treatment date.
  To handle the missing data, if a participant had at least 4 non-missing daily scores within the 7 days prior to a study visit, the weekly score was calculated as the sum of the available scores in that week, divided by the number of days with daily scores available, multiplied by 7. However, if there were less than 4 non-missing daily scores within the prior 7 days, then the weekly score was missing for the week.
Time Frame: Baseline, week 24
Population: All participants to whom study treatment was assigned. Only participants with at least 4 non-missing daily scores within the 7 days prior to the study visit at week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 23 | 13 | 11
Score on a scale | -20.36 (12.963) | -22.50 (13.503) | -21.26 (14.480)

2. Secondary Outcome: Change From Baseline of Weekly Urticaria Activity Score (UAS7) at Weeks 12 and 40
Description: as for outcome 1
Time Frame: Baseline, weeks 12 and 40
Population: All participants to whom study treatment was assigned. Only participants with at least 4 non-missing daily scores within the 7 days prior to the specified data points (weeks 12 and 40) were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Score on a scale
  Week 12: number analyzed (Participants) | 23 | 13 | 12
  Week 12 | -15.70 (10.867) | -18.38 (12.268) | -12.96 (13.043)
  Week 40: number analyzed (Participants) | 22 | 12 | 10
  Week 40 | -17.50 (12.619) | -15.65 (11.096) | -19.43 (17.667)

3. Secondary Outcome: Percentage of Participants With Complete Response in Weekly Urticaria Activity Score (UAS7)
Description: UAS7 is a self-reported scoring system to evaluate urticaria signs and symptoms. UAS7 is the sum of daily urticaria activity scores (UAS) over a seven-day period. The possible range of UAS7 score is 0 to 42 (0 to 6 for daily UAS x 7 days). A higher urticaria activity score indicates more severe symptoms. A complete UAS7 response is defined as UAS7=0, no wheals neither pruritus. Participants with post-baseline missing data were considered as non-responders.
Time Frame: Weeks 12, 24 and 40
Population: All participants to whom study treatment was assigned. Participants with post-baseline missing data were considered as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Participants
  Week 12 | 4 | 5 | 2
  Week 24 | 8 | 8 | 4
  Week 40 | 3 | 2 | 4

4. Secondary Outcome: Change From Baseline of Weekly Itch Severity Score (ISS7)
Description: ISS7 is the sum of daily Itch Severity Score (ISS) over a seven-day period. The possible range of ISS7 score is 0-21 (0-3 for daily ISS x 7 days), where 0 is defined as complete ISS7 response (no itching) and 21 is the worst score. A negative change score from baseline indicates improvement. Baseline was calculated using data from the 7 days prior to the first treatment date.
  To handle the missing data, if a participant had at least 4 non-missing daily scores within the 7 days prior to a study visit, the weekly score was calculated as the sum of the available scores in that week, divided by the number of days with daily scores available, multiplied by 7. However, if there were less than 4 non-missing daily scores within the prior 7 days, then the weekly score was missing for the week.
Time Frame: Baseline, weeks 12, 24 and 40
Population: All participants to whom study treatment was assigned. Only participants with at least 4 non-missing daily scores within the 7 days prior to the specified data points (weeks 12, 24 and 40) were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Score on a scale
  Week 12: number analyzed (Participants) | 23 | 13 | 12
  Week 12 | -7.66 (5.824) | -7.81 (6.047) | -6.34 (6.936)
  Week 24: number analyzed (Participants) | 23 | 13 | 12
  Week 24 | -9.71 (7.049) | -9.85 (6.488) | -10.28 (7.811)
  Week 40: number analyzed (Participants) | 22 | 12 | 10
  Week 40 | -8.73 (6.656) | -6.86 (5.848) | -9.88 (8.687)

5. Secondary Outcome: Percentage of Participants With Complete Response in Weekly Itch Severity Score (ISS7)
Description: ISS7 is the sum of daily Itch Severity Score (ISS) over a seven-day period. The possible range of ISS7 score is 0-21 (0-3 for daily ISS x 7 days), where 0 is defined as complete ISS7 response (no itching) and 21 is the worst score. Participants with post-baseline missing data were considered as non-responders.
Time Frame: Weeks 12, 24 and 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Participants
  Week 12 | 4 | 5 | 2
  Week 24 | 9 | 8 | 4
  Week 40 | 4 | 2 | 4

6. Secondary Outcome: Change From Baseline of Weekly Hives Severity Score (HSS7)
Description: HSS7 is the sum of daily Hives Severity Score (HSS) over a seven-day period. The possible range of HSS7 score is 0-21 (0-3 for daily HSS x 7 days), where 0 is defined as complete HSS7 response (no wheals) and 21 is the worst score. A negative change score from baseline indicates improvement. Baseline was calculated using data from the 7 days prior to the first treatment date.
  To handle the missing data, if a participant had at least 4 non-missing daily scores within the 7 days prior to a study visit, the weekly score was calculated as the sum of the available scores in that week, divided by the number of days with daily scores available, multiplied by 7. However, if there were less than 4 non-missing daily scores within the prior 7 days, then the weekly score was missing for the week.
Time Frame: Baseline, weeks 12, 24 and 40
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Score on a scale
  Week 12: number analyzed (Participants) | 23 | 13 | 12
  Week 12 | -8.03 (6.307) | -10.58 (7.225) | -6.62 (6.385)
  Week 24: number analyzed (Participants) | 23 | 13 | 11
  Week 24 | -10.65 (6.673) | -12.65 (7.785) | -10.98 (6.842)
  Week 40: number analyzed (Participants) | 22 | 12 | 10
  Week 40 | -8.77 (6.770) | -8.78 (6.084) | -9.55 (9.197)

7. Secondary Outcome: Percentage of Participants With Complete Response in Weekly Hives Severity Score (HSS7)
Description: HSS7 is the sum of daily Hives Severity Score (HSS) over a seven-day period. The possible range of HSS7 score is 0-21 (0-3 for daily HSS x 7 days), where 0 is defined as complete HSS7 response (no wheals) and 21 is the worst score. Participants with post-baseline missing data were considered as non-responders.
Time Frame: Weeks 12, 24 and 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Participants
  Week 12 | 6 | 6 | 2
  Week 24 | 10 | 9 | 4
  Week 40 | 5 | 2 | 5

8. Secondary Outcome: Change From Baseline of the Children Dermatology Life Quality Index (CDLQI)
Description: The children dermatology life quality index questionnaire is a 10-item dermatology- specific health-related quality of life measure designed for use in children. Participants rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives. The CDLQI total score is a sum of all 10 item responses, each individual response ranging from 0 (not at all) to 3 (very much). Total score ranges from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A negative change score from baseline indicates improvement. Baseline was defined as the last non-missing value prior to or on the first treatment date.
  To handle the missing data, if a participant had only one item missing score per visit, then it was imputed to 0 and total score was calculated accordingly. If there were 2 or more item missing scores per visit, then the total score for the visit was considered as missing.
Time Frame: Baseline, weeks 12, 24 and 40
Population: All participants to whom study treatment was assigned. Participants with 2 or more item missing scores at specified data points (weeks 12, 24 and 40) were not analyzed (total score for that data point was considered as missing).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Score on a scale
  Week 12: number analyzed (Participants) | 19 | 13 | 11
  Week 12 | -10.1 (4.88) | -6.6 (8.05) | -5.0 (6.23)
  Week 24: number analyzed (Participants) | 21 | 10 | 11
  Week 24 | -11.5 (6.85) | -8.8 (10.43) | -10.1 (6.74)
  Week 40: number analyzed (Participants) | 19 | 11 | 11
  Week 40 | -10.3 (6.86) | -5.5 (9.04) | -8.6 (8.54)

9. Secondary Outcome: Change From Baseline in Total Human Immunoglobulin E (IgE)
Description: Change from baseline in IgE (free IgE plus IgE bound to ligelizumab) at weeks 12, 24 and 40 as a pharmacodynamic measurement.
Time Frame: Baseline, weeks 12, 24 and 40
Population: All participants who received at least one dose of study treatment. Only those participants with data available for this endpoint at specified data points (weeks 12, 24 and 40) were analyzed.
Measure: Mean (Standard Deviation); unit: International units / millilitre
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
International units / millilitre
  Week 12: number analyzed (Participants) | 17 | 11 | 9
  Week 12 | 186 (160) | 245 (291) | -43.1 (56.2)
  Week 24: number analyzed (Participants) | 19 | 12 | 9
  Week 24 | 169 (126) | 328 (504) | 325 (411)
  Week 40: number analyzed (Participants) | 19 | 13 | 9
  Week 40 | 30.4 (105) | -15.6 (118) | -22.0 (93.0)

10. Secondary Outcome: Apparent Clearance (CL/F) of Ligelizumab Estimated With a PopPK Model
Description: Model-based estimate of apparent clearance (CL/F) was derived using compartmental pharmacokinetic population (PopPK) modelling using non-linear mixed effects model for ligelizumab. Apparent clearance population estimate was derived through fitting individual drug administration history and collected ligelizumab concentrations at the specified data points (listed in Time Frame).
Time Frame: Weeks 0 (baseline), 4, 8, 12, 16, 20 (all pre-dose) and weeks 24, 32 and 40
Population: All participants who received at least one dose of study treatment and provided an evaluable PK profile (at least 7 samples per patient collected). All ligelizumab concentration-time data were combined and included in the population PK analysis.
Measure: Median (Inter-Quartile Range); unit: Liters / day
Groups:
- All Participants With PK Data: Participants in the study (low dose, high dose and placebo+high dose) with available pharmacokinetic data
Arm/Group | All Participants With PK Data
Number analyzed (Participants) | 47
Liters / day | 0.66 [0.44 to 1.03]

11. Secondary Outcome: Apparent Volume of Distribution of Ligelizumab Estimated With a PopPK Model
Description: Model-based estimate of apparent volume of distribution was derived using compartmental pharmacokinetic population (PopPK) modelling using non-linear mixed effects model for ligelizumab. Apparent volume of distribution population estimate was derived through fitting individual drug administration history and collected ligelizumab concentrations at the specified data points (listed in Time Frame).
Time Frame: Weeks 0 (baseline), 4, 8, 12, 16, 20 (all pre-dose) and weeks 24, 32 and 40
Population: All participants who received at least one dose of study treatment and provided an evaluable PK profile (at least 7 samples per patient are required). All ligelizumab concentration-time data were combined and included in the population PK analysis.
Measure: Median (Inter-Quartile Range); unit: Liters
Arm/Group | All Participants With PK Data
Number analyzed (Participants) | 47
Liters | 14.5 [11.02 to 16.65]

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs, including significant changes from baseline in vital signs (blood pressure, pulse rate), electrocardiograms and laboratory values qualifying and reported as AEs. The number of participants in each category is reported in the table.
Time Frame: From the start of treatment to 20 weeks after end of treatment, assessed up to maximum duration of 40 weeks
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg
Number analyzed (Participants) | 24 | 13 | 12
Participants
  AEs | 18 | 11 | 9
  Treatment related AEs | 6 | 5 | 2
  SAEs | 1 | 0 | 1
  SAEs leading to treatment discontinuation | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start treatment to 20 weeks after end of treatment, assessed up to maximum duration of 40 weeks.
Groups:
- Total: Total
Arm/Group | Ligelizumab 24 mg | Ligelizumab 120 mg | Placebo + Ligelizumab 120 mg | Total
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/13 | 0/12 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/13 | 1/12 | 2/49
Other Adverse Events (participants affected / at risk) | 18/24 | 11/13 | 9/12 | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 24 mg (N=24) | Ligelizumab 120 mg (N=13) | Placebo + Ligelizumab 120 mg (N=12) | Total (N=49)
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 24 mg (N=24) | Ligelizumab 120 mg (N=13) | Placebo + Ligelizumab 120 mg (N=12) | Total (N=49)
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 4
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 5
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 4
Administration site erythema (General disorders and administration site conditions) | 0 | 1 | 0 | 1
Injection site erythema (General disorders and administration site conditions) | 0 | 0 | 1 | 1
Injection site pain (General disorders and administration site conditions) | 1 | 1 | 1 | 3
Injection site reaction (General disorders and administration site conditions) | 0 | 0 | 1 | 1
Pyrexia (General disorders and administration site conditions) | 2 | 2 | 0 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 1 | 2
Influenza (Infections and infestations) | 2 | 1 | 2 | 5
Nasopharyngitis (Infections and infestations) | 7 | 4 | 4 | 15
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 4
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 3
Headache (Nervous system disorders) | 5 | 1 | 4 | 10
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 2
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03437278/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03437278/SAP_001.pdf